CLINICAL TRIAL: NCT04337346
Title: Endometriosis Patients Covid 19 Anxiety
Brief Title: Evaluation of Covid 19 Anxiety in Endometriosis Patients
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Yalcin bahat, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: endocovid19
Record Dates: First submitted 2020-04-05; First posted 2020-04-07 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Endometriosis; Covid19
MeSH Terms: conditions — Endometriosis; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It is aimed to measure the general anxiety and lifestyle information of endometriosis patients about covid 19 pandemic, to evaluate anxiety levels in this period.

ELIGIBILITY:
Inclusion Criteria:

* endometriosis patients
* no psychiatric illness
* no antidepressant use

Exclusion Criteria:

* women who had not endometriosis
* no extra health conditions
* women younger than 18 and older than 45

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Evaluation of endometriosis patients anxiety and lifestyle during the covid 19 pandemic
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-04-05 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-04-25 (Actual)

PRIMARY OUTCOMES:
Covid 19 Anxiety levels in Endometriosis Patients | 20 days
  The Beck Anxiety Inventory (BAI); it measures the frequency of anxiety symptoms experienced by the patient. It consists of 21 questions in total. Each item gets an increasing score between 0-3. The total score ranges from 0 - 63. The following guidelines are recommended for the interpretation of scores: 0 -9, normal or no anxiety; 10 -18, mild to moderate anxiety; 19 -29, moderate to severe anxiety; and 30 - 63, severe anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Pinar Yalcin Bahat, Istanbul, İ̇stanbul, Turkey (Türkiye)